CLINICAL TRIAL: NCT02457338
Title: Infant Supplementation With Probiotic Bifidobacterium Longum Subsp. Infantis Study
Brief Title: Infant Microbiota and Probiotic Intake Study
Acronym: IMPRINT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Evolve BioSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 631099
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: C-section; Infants; Probiotic; B. infantis; Microbiota; Gut; Breast milk; Vaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement Group (Experimental): This group will receive probiotic B. infantis supplementation, plus standard care and lactation consultation.
  Interventions: Dietary Supplement: Bifidobacterium
- Control Group (No Intervention): This group will receive standard care plus lactation consultation only.

INTERVENTIONS:
Dietary Supplement: Bifidobacterium
  Other Names: B. infantis
  Arms: Supplement Group

SUMMARY:
The purpose of this study is to determine if supplementing healthy term infants delivered by C-section or vaginal delivery who only consume breastmilk with a probiotic for 21 consecutive days increases levels of bacteria in infants' stool.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to determine the effects of supplementing the probiotic Bifidobacterium longum subsp. infantis for the first 21 days of life in healthy term breastfed infants delivered via C-section or vaginal delivery on gut bacteria composition during, 1 week, and 1 month after supplementation compared with matched-control term infants receiving standard care. The investigators' specific aim is to compare the fecal microbiota (total B. infantis, total Bifidobacterium, total bacteria and composition of microbiota) between the supplement and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking women and their infants
* Who are pregnant in their third trimester OR have delivered by C-section or vaginal birth within the past 7 days
* Patients who live within a 20-mile radius from University of California Davis Medical Center (UCDMC) or a 20-mile radius from UC Davis Campus in Davis, California.
* Plan to exclusively breastfeed their infants for at least 3 months
* Infants: 0-7 days old, delivered by C-section or vaginal delivery, born >37 weeks gestation, without medical complications that would preclude breastfeeding or alter gut microbiota

Exclusion Criteria:

* Infants born with medical complications such as: respiratory distress syndrome, birth defects, and infection
* Infants who have taken antibiotics for more than 72 hours of life
* Infants who have consume formula feedings after day 7 of life
* Mothers and their infants who are not discharged from the hospital by day 4 of life due to complications
* Plan to administer probiotics to infants or use of probiotics other than the study supplement by infants anytime throughout the study duration
* Women who have had any breast surgery or injury within the past 5 years that would reduce the chance of successful exclusive breastfeeding
* Mothers who have a chronic metabolic disease or obesity

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2027-06-07 (Estimated)

PRIMARY OUTCOMES:
Infant fecal B. infantis | baseline, days 10, 14, 17, 21, 25, 29, 32, 40, 50, 60
  Measure the change from baseline, during supplementation, and post supplementation
Infant fecal Bifidobacterium | baseline, days 10, 14, 17, 21, 25, 29, 32, 40, 50, 60
  Measure the change from baseline, during supplementation, and post supplementation
Infant fecal total bacteria | baseline, days 10, 14, 17, 21, 25, 29, 32, 40, 50, 60
  Measure the change from baseline, during supplementation, and post supplementation
Infant fecal microbiota | baseline, days 10, 14, 17, 21, 25, 29, 32, 40, 50, 60
  Measure the change from baseline, during supplementation, and post supplementation
Incidence of Adverse Events and Treatments | Baseline-days 60
  Gastrointestinal symptoms and related symptoms (discomfort passing bowel movements, vomiting, constipation, colic or irritability) before, during and after B. infantis supplementation will be determined and reported daily by parental self-report questionnaire. General health status of the infant such as occurrence of any illness, health care visits for sickness, fever, antibiotic and medication use and parental assessments of infant's overall health.
Incidence of Adverse Events and Treatments | Months 4, 6, 8, 10, 12, 18 and 24
  Gastrointestinal symptoms and related symptoms (diarrhea, vomiting, constipation, colic, irritability) after B. infantis supplementation will be determined and reported parental self-report questionnaire. General health status of the infant such as occurrence of any illness, health care visits for sickness, fever, antibiotic and medication use and parental assessments of infant's overall health.

SECONDARY OUTCOMES:
Infant fecal bacteria oligosaccharide consumption | days 7, 14, 21, 32, 60
  Compare the oligosaccharides in human milk against the oligosaccharides in infant feces before, during, and after B. infantis supplementation by using liquid chromatography Chip-TOP mass spectrometry.
Infant fecal sialic acid concentrations | baseline, days 10, 14, 17, 21, 25, 29, 32, 40, 50, 60
  Measure the change in infant fecal sialic acid concentrations before, during, and after B. infantis supplementation in infant stool samples using enzymatic assay.
Maternal fecal B. infantis, Bifidobacterium, total bacteria, and microbiota composition | baseline, day 60
  Compare the maternal fecal B. infantis, bifidobacterium, total bacteria, and microbiota composition with changes in infant fecal microbiota
Infant weight | birth, hospital discharge, days 15, 33, 61
  Determine the change in weight across the study duration using a digital infant scale and change in gut microbiota
Fecal inflammatory mediators | Baseline-days 60
  Compare GI function between infants in the B. infantis and control groups through the measurement of fecal inflammatory mediators.
Fecal gut barrier function barrier markers | Baseline-days 60
  Compare GI function between infants in the B. infantis and control groups through the measurement of GI barrier function markers.
Fecal lipopolysaccharide | Baseline-days 60
  Compare GI function between infants in the B. infantis and control groups through the measurement of fecal lipopolysaccharide binding.
Fecal short-chain fatty acids | Baseline-days 60
  Determine the relationship between fecal microbiota composition and fecal short chain fatty acids
Fecal microbiome-Follow-up | Months 4, 6, 8, 10, 12
  next generation sequencing
Fecal B. infantis-Follow-up | Months 4, 6, 8, 10, 12
  Q Polymerase Chain Reaction (PCR)
Fecal Bifidobacterium-Follow-up | Months 4, 6, 8, 10, 12
  Q PCR

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Smilowitz, PhD, Principal Investigator — University of California, Davis; Mark Underwood, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Prior E, Santhakumaran S, Gale C, Philipps LH, Modi N, Hyde MJ. Breastfeeding after cesarean delivery: a systematic review and meta-analysis of world literature. Am J Clin Nutr. 2012 May;95(5):1113-35. doi: 10.3945/ajcn.111.030254. Epub 2012 Mar 28. PMID 22456657
- [Background] Bager P, Wohlfahrt J, Westergaard T. Caesarean delivery and risk of atopy and allergic disease: meta-analyses. Clin Exp Allergy. 2008 Apr;38(4):634-42. doi: 10.1111/j.1365-2222.2008.02939.x. Epub 2008 Feb 11. PMID 18266879
- [Background] Pei Z, Heinrich J, Fuertes E, Flexeder C, Hoffmann B, Lehmann I, Schaaf B, von Berg A, Koletzko S; Influences of Lifestyle-Related Factors on the Immune System and the Development of Allergies in Childhood plus Air Pollution and Genetics (LISAplus) Study Group. Cesarean delivery and risk of childhood obesity. J Pediatr. 2014 May;164(5):1068-1073.e2. doi: 10.1016/j.jpeds.2013.12.044. Epub 2014 Feb 5. PMID 24508442
- [Background] Bager P, Simonsen J, Nielsen NM, Frisch M. Cesarean section and offspring's risk of inflammatory bowel disease: a national cohort study. Inflamm Bowel Dis. 2012 May;18(5):857-62. doi: 10.1002/ibd.21805. Epub 2011 Jul 7. PMID 21739532
- [Background] Garrido D, Barile D, Mills DA. A molecular basis for bifidobacterial enrichment in the infant gastrointestinal tract. Adv Nutr. 2012 May 1;3(3):415S-21S. doi: 10.3945/an.111.001586. PMID 22585920
- [Background] Garrido D, Dallas DC, Mills DA. Consumption of human milk glycoconjugates by infant-associated bifidobacteria: mechanisms and implications. Microbiology (Reading). 2013 Apr;159(Pt 4):649-664. doi: 10.1099/mic.0.064113-0. Epub 2013 Mar 4. PMID 23460033
- [Background] Garrido D, Kim JH, German JB, Raybould HE, Mills DA. Oligosaccharide binding proteins from Bifidobacterium longum subsp. infantis reveal a preference for host glycans. PLoS One. 2011 Mar 15;6(3):e17315. doi: 10.1371/journal.pone.0017315. PMID 21423604
- [Background] Garrido D, Nwosu C, Ruiz-Moyano S, Aldredge D, German JB, Lebrilla CB, Mills DA. Endo-beta-N-acetylglucosaminidases from infant gut-associated bifidobacteria release complex N-glycans from human milk glycoproteins. Mol Cell Proteomics. 2012 Sep;11(9):775-85. doi: 10.1074/mcp.M112.018119. Epub 2012 Jun 27. PMID 22745059
- [Background] Garrido D, Ruiz-Moyano S, Jimenez-Espinoza R, Eom HJ, Block DE, Mills DA. Utilization of galactooligosaccharides by Bifidobacterium longum subsp. infantis isolates. Food Microbiol. 2013 Apr;33(2):262-70. doi: 10.1016/j.fm.2012.10.003. Epub 2012 Oct 22. PMID 23200660
- [Background] Ruiz-Moyano S, Totten SM, Garrido DA, Smilowitz JT, German JB, Lebrilla CB, Mills DA. Variation in consumption of human milk oligosaccharides by infant gut-associated strains of Bifidobacterium breve. Appl Environ Microbiol. 2013 Oct;79(19):6040-9. doi: 10.1128/AEM.01843-13. Epub 2013 Jul 26. PMID 23892749
- [Background] Underwood MA, Kalanetra KM, Bokulich NA, Lewis ZT, Mirmiran M, Tancredi DJ, Mills DA. A comparison of two probiotic strains of bifidobacteria in premature infants. J Pediatr. 2013 Dec;163(6):1585-1591.e9. doi: 10.1016/j.jpeds.2013.07.017. Epub 2013 Aug 29. PMID 23993139
- [Background] Underwood MA, Kalanetra KM, Bokulich NA, Mirmiran M, Barile D, Tancredi DJ, German JB, Lebrilla CB, Mills DA. Prebiotic oligosaccharides in premature infants. J Pediatr Gastroenterol Nutr. 2014 Mar;58(3):352-60. doi: 10.1097/MPG.0000000000000211. PMID 24135979
- [Background] Smilowitz JT, Lebrilla CB, Mills DA, German JB, Freeman SL. Breast milk oligosaccharides: structure-function relationships in the neonate. Annu Rev Nutr. 2014;34:143-69. doi: 10.1146/annurev-nutr-071813-105721. Epub 2014 May 15. PMID 24850388
- [Background] Sela DA. Bifidobacterial utilization of human milk oligosaccharides. Int J Food Microbiol. 2011 Sep 1;149(1):58-64. doi: 10.1016/j.ijfoodmicro.2011.01.025. Epub 2011 Jan 26. PMID 21342711
- [Background] Sela DA, Chapman J, Adeuya A, Kim JH, Chen F, Whitehead TR, Lapidus A, Rokhsar DS, Lebrilla CB, German JB, Price NP, Richardson PM, Mills DA. The genome sequence of Bifidobacterium longum subsp. infantis reveals adaptations for milk utilization within the infant microbiome. Proc Natl Acad Sci U S A. 2008 Dec 2;105(48):18964-9. doi: 10.1073/pnas.0809584105. Epub 2008 Nov 24. PMID 19033196
- [Background] Sela DA, Garrido D, Lerno L, Wu S, Tan K, Eom HJ, Joachimiak A, Lebrilla CB, Mills DA. Bifidobacterium longum subsp. infantis ATCC 15697 alpha-fucosidases are active on fucosylated human milk oligosaccharides. Appl Environ Microbiol. 2012 Feb;78(3):795-803. doi: 10.1128/AEM.06762-11. Epub 2011 Dec 2. PMID 22138995
- [Background] Sela DA, Li Y, Lerno L, Wu S, Marcobal AM, German JB, Chen X, Lebrilla CB, Mills DA. An infant-associated bacterial commensal utilizes breast milk sialyloligosaccharides. J Biol Chem. 2011 Apr 8;286(14):11909-18. doi: 10.1074/jbc.M110.193359. Epub 2011 Feb 2. PMID 21288901
- [Background] Sela DA, Mills DA. Nursing our microbiota: molecular linkages between bifidobacteria and milk oligosaccharides. Trends Microbiol. 2010 Jul;18(7):298-307. doi: 10.1016/j.tim.2010.03.008. Epub 2010 Apr 19. PMID 20409714
- [Background] LoCascio RG, Ninonuevo MR, Freeman SL, Sela DA, Grimm R, Lebrilla CB, Mills DA, German JB. Glycoprofiling of bifidobacterial consumption of human milk oligosaccharides demonstrates strain specific, preferential consumption of small chain glycans secreted in early human lactation. J Agric Food Chem. 2007 Oct 31;55(22):8914-9. doi: 10.1021/jf0710480. Epub 2007 Oct 5. PMID 17915960
- [Background] LoCascio RG, Desai P, Sela DA, Weimer B, Mills DA. Broad conservation of milk utilization genes in Bifidobacterium longum subsp. infantis as revealed by comparative genomic hybridization. Appl Environ Microbiol. 2010 Nov;76(22):7373-81. doi: 10.1128/AEM.00675-10. Epub 2010 Aug 27. PMID 20802066
- [Background] Dominguez-Bello MG, Costello EK, Contreras M, Magris M, Hidalgo G, Fierer N, Knight R. Delivery mode shapes the acquisition and structure of the initial microbiota across multiple body habitats in newborns. Proc Natl Acad Sci U S A. 2010 Jun 29;107(26):11971-5. doi: 10.1073/pnas.1002601107. Epub 2010 Jun 21. PMID 20566857
- [Background] Penders J, Gerhold K, Stobberingh EE, Thijs C, Zimmermann K, Lau S, Hamelmann E. Establishment of the intestinal microbiota and its role for atopic dermatitis in early childhood. J Allergy Clin Immunol. 2013 Sep;132(3):601-607.e8. doi: 10.1016/j.jaci.2013.05.043. Epub 2013 Jul 27. PMID 23900058
- [Background] Penders J, Thijs C, Vink C, Stelma FF, Snijders B, Kummeling I, van den Brandt PA, Stobberingh EE. Factors influencing the composition of the intestinal microbiota in early infancy. Pediatrics. 2006 Aug;118(2):511-21. doi: 10.1542/peds.2005-2824. PMID 16882802
- [Result] Henrick BM, Hutton AA, Palumbo MC, Casaburi G, Mitchell RD, Underwood MA, Smilowitz JT, Frese SA. Elevated Fecal pH Indicates a Profound Change in the Breastfed Infant Gut Microbiome Due to Reduction of Bifidobacterium over the Past Century. mSphere. 2018 Mar 7;3(2):e00041-18. doi: 10.1128/mSphere.00041-18. eCollection 2018 Mar-Apr. PMID 29564397
- [Result] Casaburi et al., Colonization of breastfed infants by Bifidobacterium longum subsp. infantis EVC001 reduces virulence gene abundance
- [Result] Karav S, Casaburi G, Frese SA. Reduced colonic mucin degradation in breastfed infants colonized by Bifidobacterium longum subsp. infantis EVC001. FEBS Open Bio. 2018 Sep 17;8(10):1649-1657. doi: 10.1002/2211-5463.12516. eCollection 2018 Oct. PMID 30338216
- [Result] Frese SA, Hutton AA, Contreras LN, Shaw CA, Palumbo MC, Casaburi G, Xu G, Davis JCC, Lebrilla CB, Henrick BM, Freeman SL, Barile D, German JB, Mills DA, Smilowitz JT, Underwood MA. Persistence of Supplemented Bifidobacterium longum subsp. infantis EVC001 in Breastfed Infants. mSphere. 2017 Dec 6;2(6):e00501-17. doi: 10.1128/mSphere.00501-17. eCollection 2017 Nov-Dec. PMID 29242832
- [Result] Smilowitz JT, Moya J, Breck MA, Cook C, Fineberg A, Angkustsiri K, Underwood MA. Erratum to: Safety and tolerability of Bifidobacterium longum subspecies infantis EVC001 supplementation in healthy term breastfed infants: a phase I clinical trial. BMC Pediatr. 2017 Aug 15;17(1):180. doi: 10.1186/s12887-017-0932-7. No abstract available. PMID 28810848
- [Derived] Casaburi G, Duar RM, Vance DP, Mitchell R, Contreras L, Frese SA, Smilowitz JT, Underwood MA. Early-life gut microbiome modulation reduces the abundance of antibiotic-resistant bacteria. Antimicrob Resist Infect Control. 2019 Aug 14;8:131. doi: 10.1186/s13756-019-0583-6. eCollection 2019. PMID 31423298
- [Derived] Smilowitz JT, Moya J, Breck MA, Cook C, Fineberg A, Angkustsiri K, Underwood MA. Safety and tolerability of Bifidobacterium longum subspecies infantis EVC001 supplementation in healthy term breastfed infants: a phase I clinical trial. BMC Pediatr. 2017 May 30;17(1):133. doi: 10.1186/s12887-017-0886-9. PMID 28558732